CLINICAL TRIAL: NCT02843373
Title: Longitudinal, Prospective Study to Examine the Brain-based Biomarkers of Response to Transcranial Magnetic Stimulation Treatment in Major Depressive Disorder
Brief Title: Brain-Based Biomarkers in Response to TMS in MDD
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Corey Keller, Assistant Professor of Psychiatry and Behavioral Sciences, Stanford University
Other Study IDs: IRB-25948
Record Dates: First submitted 2016-07-20; First posted 2016-07-25 (Estimated); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Major Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rTMS: rTMS will be delivered for 20 sessions over 4 weeks. Active 10 Hz rTMS will be delivered to the left DLPFC as assessed by either the 5cm rule or F3 site. Daily treatment regiments will last 36.5 minutes and rTMS will be delivered at 120% of the participant's motor threshold. Participants will be monitored during the rTMS sessions for adverse events and/or side effects.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS

SUMMARY:
The overarching goal of this research program is to elucidate causal and directional neural network- level abnormalities in depression, and how they are modulated by an individually-tailored, circuit-directed intervention. By using concurrent TMS and EEG, the investigators can overcome a major limitation of EEG - the inability to demonstrate causality. Here, we plan to recruit patients with medication-resistant depression undergoing rTMS treatment. At multiple time points, we will perform TMS-EEG to investigate the excitability and connectivity profiles of brain networks and how they are modulated during treatment. This study aims to provide objective brain network measures that can predict and track clinical response to TMS treatment. Findings from this study will be utilized to develop a novel, personalized treatment protocol based on individual brain networks.

DETAILED DESCRIPTION:
Goals of the study are as follows:

* To evaluate the ability to predict and track brain network changes during TMS treatment for medication-resistant depression.
* To develop quantitative tools that measure the connectivity and excitability of the brain using resting and single pulse TMS-EEG.
* To determine the feasibility of recording EEG biomarkers in the clinic without disrupting clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 to 60
* Medication-resistant depression as assessed by psychiatrist
* Must comprehend English well to ensure adequate comprehension of the EEG and TMS instructions, and of clinical scales
* Has failed >1 previous adequate antidepressant medication trials
* Right-handed
* No current or history of neurological disorders
* No seizure disorder or risk of seizures
* No use of PRN medication within 48 hours of the scheduled study appointment

Exclusion Criteria:

* Any unstable medical condition, any significant CNS neurological condition such as stroke, seizure, tumor, hemorrhage, multiple sclerosis, etc
* Current electroconvulsive therapy (ECT) or prior treatment failure with ECT
* Currently pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community care clinic
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-03; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
TMS-EEG | Up to 3 months
  From pre- to post-treatment, improvement will be based on enhanced excitability and connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Corey Keller, MD PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No